CLINICAL TRIAL: NCT05522049
Title: Videolaryngoscopy-guided Intubation Using Macintosh Versus Hyperangulated Blades in Patients With Expected Difficult Intubation Undergoing Ear, Nose and Throat Surgery or Maxillofacial Surgery a Randomized Controlled Trial
Brief Title: Videolaryngoscopic Intubation Using Macintosh vs.Hyperangulated Blades in Patients With Expected Difficult Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-100868-BO-ff
Record Dates: First submitted 2022-08-22; First posted 2022-08-30 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Intubation; Difficult or Failed; Videolaryngoscopy; General Anesthesia
Keywords: Airway management; Hyperangulated blade; Macintosh blade

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Tracheal intubation facilitated by a hyperangulated videolaryngoscope (C-MAC D-Blade)
  Interventions: Device: hyperangulated videolaryngoscope
- Control group (Active Comparator): Tracheal intubation facilitated by a videolaryngoscope with a Macintosh type blade (C-MAC)
  Interventions: Device: Macintosh videolaryngoscope

INTERVENTIONS:
Device: hyperangulated videolaryngoscope — Intubation using a hyperangulated videolaryngoscope
  Other Names: C-MAC D-Blade; Storz
  Arms: Intervention group
Device: Macintosh videolaryngoscope — Intubation using a Macintosh videolaryngoscope
  Other Names: C-MAC; Storz
  Arms: Control group

SUMMARY:
Videolaryngoscopy-guided intubation has become widespread as a means of preventing major complications relating to airway management by improving the glottic view, increasing the first attempt success rate, likely reduce rates of hypoxemic events, while reducing the rate of airway trauma. However, as randomized controlled studies in patients with anticipated difficult intubation undergoing ear nose and throat (ENT) or oral and maxillofacial (OMF) surgery are lacking, it is still unknown if hyperangulated blades improve glottic view and if their use translates into faster intubation. The primary aim of this randomized controlled trial is to compare the percentage of glottic opening (POGO) between hyperangulated blades and Macintosh blades in patients with expected difficult intubation undergoing ENT or OMF surgery who require transoral tracheal intubation. Secondary aims are to compare secondary outcome measures such as time variables, indicators for difficult and successful intubation, number of attempts, view conditions, difficult airway classifications and adverse events between both blade types.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring general anesthesia with transoral tracheal intubation for elective ear, nose and throat or maxillofacial surgery
* Expected difficult intubation
* Age ≥ 18

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Planned awake tracheal intubation (without deep anesthesia or neuromuscular blocking agents)
* Required transnasal tracheal intubation (e.g. for surgical reasons)
* Special tubes required for surgical reasons ( e.g. double lumen tube)
* Denial of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of glottic opening (POGO) | 1 hour
  Grading of the best view obtained during laryngoscopy (%)

SECONDARY OUTCOMES:
Time to successful tracheal intubation (seconds) | 1 hour
  Recorded during airway management
Time to successful first attempt intubation (seconds) | 1 hour
  Recorded during airway management
Cormack-Lehane grade | 1 hour
  Grading of the best view obtained during laryngoscopy (I [best] to IV [worst])
Impaired view (vocal cords cannot be visualized by laryngoscopy) | 1 hour
  Number of participants with impaired view observed during airway management
Difficult laryngoscopy | 1 hour
  Number of participants with difficult laryngoscopy as defined in current guidelines
Difficult intubation | 1 hour
  Number of participants with difficult tracheal intubation as defined in current guidelines
Transition to a different tracheal intubation technique | 1 hour
  Number of participants in whom the airway operator decided to convert to an alternative intubation technique
Tracheal introducer | 1 hour
  Number of participants in whom the airway operator decided to use a tracheal introducer
Successful first attempt | 1 hour
  Number of participants with successful tracheal intubation with only one attempt
Overall success of intubation | 1 hour
  Number of participants with successful tracheal intubation regardless of the the number of attempts
Difficulty of videolaryngoscope-guided intubation | 1 hour
  VIDIAC (Videolaryngoscopic Intubation and Difficult Airway Classification) Score from -1 (best) to 5 (worst)
Number of intubation attempts | 1 hour
  Observed during airway management
Number of laryngoscopy attempts | 1 hour
  Observed during airway management
Airway related adverse events | 1 hour
  Number of participants with airway related adverse events observed during airway management
Hypoxaemia | 1 hour
  Number of participants with a drop in peripheral oxygen saturation during airway management
Hypotension | 1 hour
  Number of participants with hypotension observed during airway management

CONTACTS AND LOCATIONS:
Overall Officials: Martin Petzoldt, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany